CLINICAL TRIAL: NCT02087956
Title: Patient Priorities and Community Context: Navigation for Disadvantaged Women With Depression
Brief Title: Realizing Opportunities for Self Empowerment
Acronym: ROSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Ellen Poleshuck, Director, Women's Behavioral Health Service; Associate Professor, Departments of Psychiatry and Obstetrics & Gynecology, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AD-12-11-4261
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Results first posted 2019-01-07 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Depression
Keywords: Women; Depression; Socioeconomically Disadvantaged; Navigation
MeSH Terms: conditions — Depression | interventions — Referral and Consultation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Personalized Support for Progress (PSP) (Active Comparator): In Personalized Support for Progress (PSP), patients meet with a navigator to prioritize their concerns using a decision aid, develop a plan based on their identified priorities, and execute the plan.
  Interventions: Behavioral: Navigation
- Enhanced Screening and Referral (ESR) (Active Comparator): (ESR)- participant will receive personal report of their current needs and list of resources available in the community.
  Interventions: Behavioral: Enhanced Screening and Referral

INTERVENTIONS:
Behavioral: Navigation — The navigator provides up to 4 months outreach and support to implement the personal care plan. Patients determine the preferred frequency and type of contact with the navigator. . At the end of the four months, the patient and navigator will review the personal care plan, and the navigator will work with the patient as to how she can continue progress through accessing other supports and resources as needed.
  Other Names: mentoring
  Arms: Personalized Support for Progress (PSP)
Behavioral: Enhanced Screening and Referral — Patients assigned to ESR will be provided with a print-out of their Promote-W comprehensive health screening results. More specifically, they will receive a list of concerns they endorsed plus a resource list of locations where they can obtain assistance with those issues, which are largely free.
  Other Names: Comprehensise health result screening
  Arms: Enhanced Screening and Referral (ESR)

SUMMARY:
The purpose of this study is to determine whether priority-based patient navigation will improve patient satisfaction, quality of life (QOL), and depression when compared to screening-and-referral for socioeconomically disadvantaged women's health patients with depression. The investigators goal is to establish patient-driven, effective, generalizable, and disseminable interventions to reduce depression-related disparities and improve outcomes.

DETAILED DESCRIPTION:
* In this comparative effectiveness study, 200 participants who are patients at the University of Rochester Women's Health Practice or Highland Woman's Health and report significant depressive symptoms will be randomized to either PSP (Personal Support for Progress) or ESR (Enhanced Screening and Referral). Participants assigned to PSP will work with a patient navigator to prioritize their concerns, develop a personalized care plan, and implement their plan. Participants assigned to ESR will receive a personalized report of community resources that may be helpful for their identified needs.
* The investigators will use a simple 1:1 randomized design with treatment assignment being conducted using a random number generator. All analyses will follow an intent-to-treat protocol, such that all participants randomized will be followed for data collection and analyzed according to her randomized condition
* Each participant will be assessed 4 times for outcome changes: at baseline, post treatment (4 months), and two follow up ( at 7 and 10 months).
* Assessments are self report on iPads and they are linked directly to a Red Cap database.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with depression (PHQ9 score 10 or higher)
* Patient of University of Rochester Women's Health Practice or Highland Women's Health
* Monroe County resident
* English speaking

Exclusion Criteria:

* Currently receiving case management services
* In need of acute psychiatric services
* Unable to commit to the duration of the project

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2014-01; Primary Completion 2016-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Poleshuck, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Women Health Practice, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Personalized Support for Progress (PSP) | Enhanced Screening and Referral (ESR)
Started | 111 | 112
Completed | 105 | 107
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Population: We enrolled 223 participants into this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Personalized Support for Progress (PSP) | Enhanced Screening and Referral (ESR) | Total
Number analyzed (Participants) | 111 | 112 | 223
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.7 (8.8) | 30.5 (10.1) | 30.1 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 112 | 223
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Our demographic measure included both race and ethnicity (Hispanic/Latina) in one category. Population: Our sample doesn't add up to 100% because our participant could check "all that apply" for race/ethnicity.
  Participants
    AA/Black | 69 | 68 | 137
    White/Caucasian | 26 | 27 | 53
    Hispanic/Latina | 19 | 24 | 43
    Other (Native American, Asian, Hawaiian) | 4 | 8 | 12
    Biracial/More than one race | 7 | 11 | 18
Region of Enrollment [Number; unit: participants]
  United States | 111 | 112 | 223

OUTCOME MEASURES:

1. Primary Outcome: Patient Quality of Life
Description: We will use the WHOQOL-BREF measure. The WHOQOL-bref contains 26 items; the first two questions evaluate self-perceived quality of life and satisfaction with health.The remaining 24 questions represent four domains: physical, psychological, social relationships and environment.
  The WHOQOL-bref contains five Likert style response scales: "very poor to very good" (evaluation scale), "very dissatisfied to very satisfied" (evaluation scale), "none to extremely" (intensity scale), "none to complete" (capacity scale) and "never to always" (frequency scale).The mean score in each domain indicates the individual's perception of their satisfaction with each aspect of their life, relating it with quality of life. The higher the score, the better this is perceived to be. Total score was computed by summing all 26 items. The possible range is from 26 to 130.
Time Frame: Post treatment (4 months after enrollment)
Population: Results are presented for WHO-QOL total score. We had attrition of about 5% throughout the study, therefore number of analyzed at post treatment differs from initial number of participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Personalized Support for Progress (PSP) | Enhanced Screening and Referral (ESR)
Number analyzed (Participants) | 111 | 112
units on a scale
  baseline | 79.51 (13.82) | 76.91 (13.70)
  post treatment: number analyzed (Participants) | 105 | 107
  post treatment | 82.70 (14.14) | 78.85 (15.57)

2. Primary Outcome: Depression Change Outcome Measure
Description: Depression was measured by PHQ-9, a screen for major depressive disorder with good discriminant validity and sensitivity to change validated in Ob/Gyn settings, and with pregnant and postpartum women, and with women of color. Scale ranges 0-27. Higher the score, higher severity of depression and cutpoints of 5, 10, 15 and 20 representing mild, moderate, moderately severe and severe levels of depressive symptoms.
Time Frame: baseline, post treatment (4 months after enrollment), 3 months and 6 months follow up (7 and 10 months after enrollment)
Population: We had 5% attrition throughout the study, therefore number of subjects differ at each assessment point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Personalized Support for Progress (PSP) | Enhanced Screening and Referral (ESR)
Number analyzed (Participants) | 111 | 112
units on a scale
  baseline | 13.92 (3.78) | 14.74 (4.21)
  post treatment: number analyzed (Participants) | 105 | 107
  post treatment | 10.61 (6.43) | 12.58 (6.56)
  3 months follow-up: number analyzed (Participants) | 105 | 106
  3 months follow-up | 10.14 (6.19) | 11.39 (6.45)
  6 months follow-up: number analyzed (Participants) | 105 | 105
  6 months follow-up | 10.21 (6.27) | 10.36 (6.40)

3. Primary Outcome: Client Satisfaction Questionnaire- 8 Items
Description: The Client Satisfaction Questionnaire (CSQ-8) is an 8-item self-report instrument to assess subjective satisfaction with treatment which was administered to all participants post-treatment We analyzed 4 items: CSQ1: "How would you rate the quality of service you have received?", CSQ 3: "To what extent has our program met your needs?", CSQ 6: "Have the services you received helped you to deal more effectively with your problems?" and CSQ 7: "In an overall, general sense, how satisfied are you with the service you have received?" (1 = Excellent, 2 = Good, 3 = Fair, 4 = Poor). We are reporting on CSQ 1 outcome.
Time Frame: Post treatment- 4 months after enrollment, 3 and 6 months follow-up (7 and 10 months after the enrollment)
Population: We had attrition of about 5% throughout the study, therefor number of analyzed at post treatment differs from initial number of participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enhanced Screening and Referral (ESR) | Personalized Support for Progress (PSP)
Number analyzed (Participants) | 106 | 105
units on a scale
  CSQ 1. post treatment | 1.57 (0.65) | 1.43 (0.65)
  CSQ 1. 3 months follow-up | 1.72 (0.70) | 1.50 (0.64)
  CSQ 1. 6 months follow-up: number analyzed (Participants) | 105 | 104
  CSQ 1. 6 months follow-up | 1.63 (0.75) | 1.41 (0.62)

4. Secondary Outcome: Domestic Violence (Feldhaus)
Description: Feldhaus Partner Violence Screen is 3 items measure assessing physical abuse by partner in the past year. Scale range: 0-3; higher the score higher frequency of physical abuse.
Time Frame: baseline, post treatment (4 months after enrollment), 3 and 6 months follow-up (7 and 10 months after enrollment)
Population: We had attrition of 5% throughout the study; additionally we had some missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Personalized Support for Progress (PSP) | Enhanced Screening and Referral (ESR)
Number analyzed (Participants) | 108 | 109
units on a scale
  DV_baseline | 0.29 (0.45) | 0.23 (0.42)
  DV_post treatment: number analyzed (Participants) | 104 | 106
  DV_post treatment | 0.17 (0.38) | 0.26 (0.44)
  DV_3 months follow-up: number analyzed (Participants) | 104 | 106
  DV_3 months follow-up | 0.17 (0.38) | 0.23 (0.42)
  DV_6 months follow-up: number analyzed (Participants) | 104 | 105
  DV_6 months follow-up | 0.11 (0.31) | 0.20 (0.40)

ADVERSE EVENTS:
Groups:
- Personalized Support for Progress (PSP): In Personalized Support for Progress (PSP), patients meet with a navigator to prioritize their concerns using a decision aid, develop a plan based on their identified priorities, and execute the plan.
  Navigation: The navigator provides up to 4 months outreach and support to implement the personal care plan. Patients determine the preferred frequency and type of contact with the navigator. At the end of the four months, the patient and navigator will review the personal care plan, and the navigator will work with the patient as to how she can continue progress through accessing other supports and resources as needed.
- Enhanced Screening and Referral (ESR): Enhanced Screen and Referral (ESR)- participant will receive personal report of their current needs and list of resources available in the community.
  Enhanced Screening and Referral: Patients assigned to ESR will be provided with a print-out of their Promote-W comprehensive health screening results. More specifically, they will receive a list of concerns they endorsed plus a resource list of locations where they can obtain assistance with those issues, which are largely free.
Arm/Group | Personalized Support for Progress (PSP) | Enhanced Screening and Referral (ESR)
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/112
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/112
Other Adverse Events (participants affected / at risk) | 0/111 | 0/112

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No